CLINICAL TRIAL: NCT06395363
Title: Evaluation of the Functional Outcomes of Surgical Treatment in Displaced, Closed, and Isolated Distal Clavicle Fractures in Adults, A Comparative Retrospective Study
Brief Title: Evaluation of the Functional Outcomes of Surgical Treatment in Displaced, Closed, and Isolated Distal Clavicle Fractures in Adults
Acronym: clavicle_fruc
Status: Completed | Type: Observational
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Other Study IDs: Tishreen_ Clavical fructures; 15 (Registry Identifier: Tishreen_University)
Record Dates: First submitted 2024-04-25; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Clavicle Fracture
Keywords: Distal clavicle fractures; TBW; Hook plate; functional outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tension Band Wiring (TBW) group: Patients had The fixation method that involved trans-articular fixation through the acromioclavicular joint, supplemented with an additional cerclage wire tension band for enhanced stability. Following surgery, the operated shoulder was supported with a triangular sling for a period of 4 to 6 weeks. Gentle mobilization was permitted once pain subsided, although full range of motion was limited due to pin impingement until implant removal.
  Interventions: Procedure: fixation method
- In the Hook plate group: Patients had The fixation method that involved creating a tunnel in the sub-acromial space posterior to the acromioclavicular joint and inserting the hook into this tunnel. If necessary, the plate was contoured to match the clavicle's shape, with careful consideration given to the appropriate depth of the hook. Dynamic compression was utilized to secure the plate in place. Following surgery, the shoulder was supported with a triangular sling for a period ranging from 2 to 4 weeks. Mobilization commenced at the earliest opportunity, typically resulting in full range of motion within three to four weeks. It is worth mentioning that across both groups, heavy manual labor was prohibited until evidence of solid fracture union was observed.
  Interventions: Procedure: fixation method

INTERVENTIONS:
Procedure: fixation method — The fixation methods were either involved trans-articular fixation through the acromioclavicular joint, supplemented with an additional cerclage wire tension band for enhanced stability. Or, creating a tunnel in the sub-acromial space posterior to the acromioclavicular joint and inserting the hook into this tunnel.

SUMMARY:
Clavicle fractures are common among young people, generally as a consequence of car accidents, bike falls, and contact sports injuries. 15-20% of all clavicle fractures involve the lateral end of the bone. Thus, the distal clavicle fractures, in particular, have a high nonunion rate ranging from 21-33% when treated non-operatively, underscoring the usual advice for operative treatment. While significant research has been conducted on clavicle fractures and their treatment options, no definitive guidelines or optimal approaches have been established. Hence, this study aimed at assessing the clinical and radiological results of the two highly used surgical techniques, the Tension Band Wiring (TBW) and Hook plate ones, in addition to investigating the associated functional recovery and outcomes.

DETAILED DESCRIPTION:
Clavicle fractures are common among young people, generally as a consequence of car accidents, bike falls, and contact sports injuries. 15-20% of all clavicle fractures involve the lateral end of the bone. Thus, the distal clavicle fractures, in particular, have a high nonunion rate ranging from 21-33% when treated non-operatively, underscoring the usual advice for operative treatment. While significant research has been conducted on clavicle fractures and their treatment options, no definitive guidelines or optimal approaches have been established. Hence, this study aimed to assess the clinical and radiological results of the two highly used surgical techniques, Tension Band Wiring (TBW) and Hook plate ones, in addition to investigating the associated functional recovery and outcomes.

Between August 2019 and 2022, An analytical retrospective comparative study was done on 38 patients (20 TBW and 18 Hook plate) diagnosed with a fracture of the lateral third of clavicle (Neer 2) and followed up for more than 12 months at Tishreen University Hospital, Lattakia, Syria.

This research study included patients who met the following criteria: Patients with unstable distal third clavicle fracture (Neer type 2), aged between 18 and 65 years old. Nevertheless, Patients who had open fractures, pathological fractures, fractures associated with brachial plexus or pulmonary or vascular injury, acromioclavicular joint disruption, and musculoskeletal disease that affects the joint, were excluded.

Preoperative shoulder x-rays in AP with (10-15) ° cephalic tilt (ZANCA View) and axillary view were taken. In addition, Basic lab tests were done for all patients on admission. this study used A.O Hook plate with (4-7) holes, (3.5) mm screws, and (12.15.18) mm of hook depth, 2 Kirschner-wires of (2.0) mm, and a stainless steel wire of (18) gauge in the TBW technique.

Furthermore, Radiological assessment was performed immediately after surgery, followed by evaluations at 3, 6, 12, and 24-week intervals to monitor healing progress and implant positioning. Recorded complications included infection, non-union, mal-union, pin migration, hardware impingement, and stiffness. The outcome was assessed based on union status, time to fracture union, shoulder joint range of motion, ability to perform daily activities and return to pre-injury status

ELIGIBILITY:
Inclusion Criteria:

* Patients with unstable distal third clavicle fracture (Neer type 2)
* Patients aged between 18 and 65 years old

Exclusion Criteria:

* Patient who had open fractures, pathological fractures, fractures associated with brachial plexus or pulmonary or vascular injury, acromioclavicular joint disruption, and musculoskeletal disease that affects the joint

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is a comparative retrospective study of 38 patients who had unstable distal clavicle fracture (Neer 2) featured in Figure 1. treated either with TBW technique (Figure 3 and 4) or A.O Hook plate fixation (Fugure.2), and presented to the orthopedic department of Tishreen University Hospital, in Lattakia, Syria, between August 30, 2019 and August 30, 2022.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
The Rate of Wound infection | Estimated time is up to 6 weeks, follow-up visits typically at 2 weeks, 4 weeks, and 6 weeks post-surgery.
  Wound infection refers to the occurrence of microbial contamination or colonization leading to clinical signs and symptoms of infection at the surgical site. It encompasses various types of infections, including superficial, deep, and organ/space surgical site infections, as defined by the Centers for Disease Control and Prevention (CDC) criteria.
The Rate of wire migration | Up to 12 months, Regular monitoring of wire stability and migration during scheduled follow-up visits, typically conducted monthly for the duration of the study.
  The rate of wire migration refers to the occurrence of movement or displacement of wires used in surgical procedures, particularly those intended for fixation or support, Wire migration can lead to various complications depending on the location and purpose of the wire, including malpositioning, tissue damage, or loss of efficacy in providing support or stabilization.
The incidence of sub-acromial impingement | Continued monitoring of shoulder function and pain at intermediate time points during the study, up to 12 months post-treatment,
  Sub-acromial impingement syndrome is a common shoulder disorder characterized by compression or irritation of the structures located beneath the acromion, including the rotator cuff tendons and sub-acromial bursa.
The Rate of Skin erosion | Continued monitoring immediate post-intervention period up to 12 months post operatively.
  Skin erosion refers to the gradual wearing away or breakdown of the skin surface, leading to the exposure of underlying tissues.skin erosion may occur as a result of various factors, including the type of medical device or implant used, repeated friction or pressure on the skin, or underlying infection. Monitoring skin erosion is important as it can indicate potential complications related to the intervention, such as device failure, tissue irritation, or infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Tishreen University, Latakia, Syria

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT06395363/Prot_SAP_000.pdf